CLINICAL TRIAL: NCT01733173
Title: Pilot Study: Functional Imaging of Cerebellar Mutism Syndrome
Brief Title: Functional Imaging of Cerebellar Mutism Syndrome
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 12-121
Record Dates: First submitted 2012-11-20; First posted 2012-11-26 (Estimated); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Brain Mass
Keywords: mass in posterior fossa; benign; malignant; surgical resection; MRI; fMRI; DTI; 12-121
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; Diffusion Tensor Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- mass in posterior fossa, either benign or malignant: A pilot study will be performed. We will perform fMRI and DTI in children before and after surgery for posterior fossa brain tumors. Each subject will receive the standard of care for their brain tumors in terms of surgical resection, radiation therapy and/or chemotherapy.
  Interventions: Procedure: MRI with DTI and fMRI

INTERVENTIONS:
Procedure: MRI with DTI and fMRI — When possible, the subject will undergo a post operative fMRI/ DTI scan as well as clinical language testing. If the subject develops CMS, the second fMRI will be performed as soon as possible. Some subjects may be severely impaired or have difficulty performing fMRI and clinical language testing tasks. In these instances, the fMRI and language testing may not be performed, or we may choose to perform resting state or passive fMRI tasks instead.

SUMMARY:
The purpose of this study is to better understand why some children with cancer have difficulty speaking after brain surgery. Difficulty speaking may be due to known complications to the language centers in the brain. These language centers may be located in slightly different places in different people. This study will study which areas may be damaged.

ELIGIBILITY:
Inclusion Criteria:

* Subject and/or guardian is able to provide written informed consent prior to study registration
* Age ≥3 years and ≤21 years
* Newly diagnosed, untreated mass in posterior fossa, either benign or malignant
* Is being evaluated for surgical resection of the mass
* Able to perform clinical language testing in English

Exclusion Criteria:

* Claustrophobia
* Any contraindication to MRI (e.g., pacemaker, aneurysm clip, tissue expander).
* Pregnant or nursing female
* Does not speak English as a primary language (as determined by the P.I. or treating physician after discussion with a potential subject and his/her family)
* Preexisting language or developmental disorder that would limit ability to cooperate with testing (as determined by the P.I. or treating physician after interviewing potential subject and his/her family; for example, a child may be excluded if he/she has confirmed or suspected autism spectrum disorder, dysarthria, dyslexia, lisp, hypotonia, or other age inappropriate speech development)

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: MSK clinics
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2012-11; Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
investigate the feasibility of performing preoperative fMRI | 1 year
  in young children at risk for developing CMS after posterior fossa brain tumor resection. Age appropriate language functional MRI tasks targeting the cerebellar language centers will be performed in children before surgery and correlated with formal neuropsychological and language testing. The fMRI will be repeated after surgery. If ≥5 of the 7 subjects successfully complete ≥60% of the functional imaging tests, we will determine the pilot study to be successful and then pursue further study.

SECONDARY OUTCOMES:
To investigate potential changes in Diffusion Tensor Imaging (DTI) and tractography | 1 year
  in subjects who develop CMS after brain tumor resection. Injury to cerebro-cerebellar tracts such as the dentatothalamocortical tracts has been implicated in the development of CMS. We propose studying the proximity between important language white matter paths and the surgical intervention before surgery. DTI: Measurements of DTI parameters (e.g., fractional anisotropy, apparent diffusion coefficient) of cerebellar and cerebro-cerebellar white matter tracts on the preoperative scan
To investigate potential changes in DTI after posterior fossa surgery | 1 year
  that may correlate with the development of CMS. We hypothesize that measurements of water diffusion by DTI and tractography will be altered in subjects who develop CMS, even without striking anatomical changes after surgery. DTI: Measurements of DTI parameters (e.g., fractional anisotropy, apparent diffusion coefficient) of cerebellar and cerebro-cerebellar white matter tracts on the postoperative scan. The preoperative and postoperative DTI results will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Young, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/